CLINICAL TRIAL: NCT07004166
Title: Effects of TPR Technique and Z Technique on Pain and Drug Leakage in Intramuscular Injections
Brief Title: Effects of TPR and Z Techniques on Pain and Drug Leakage in Intramuscular Injections
Acronym: TPR_Z_PainLeak
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Hulya Kocyigit, Phd, Research Assitant, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15.05/2025 C
Record Dates: First submitted 2025-05-13; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Muscle Pain; Injection Site Pain
Keywords: Intramuscular Injection; Drug Leakage l; Pain; Z-Track; TPR Techniques
MeSH Terms: conditions — Myalgia; Pain

STUDY DESIGN:
Intervention Model Description: Procedure:
  Each participant will receive two injections, one into each ventrogluteal muscle. One side will be randomly assigned to the Z-track method, the other to the TPR method, using coin toss randomization. All injections will be administered by the same researcher using 3 mL of diclofenac sodium with a 21G (0.80x38 mm) needle. Injection speed will be 1 mL per 10 seconds.
  For the Z-track method, the skin will be pulled laterally by 2.5-3.5 cm before needle insertion at a 90-degree angle. After aspiration and injection, the needle will be withdrawn and the skin released immediately.
  For the TPR method, while the needle is inserted at a 90-degree angle, deep pressure will be applied to the muscle, then rapidly released to create a snapping motion that facilitates the injection. This technique relies on rapid muscle relaxation rather than needle movement by the dominant hand.
  A second blinded researcher will immediately measure leakage diameter with a millimeter ruler and evaluate
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPR (traction-pressure-release) technique (Experimental): Intervention Type: Intramuscular drug administration with TPR technique Intervention Name: Diclofenac Sodium
  TPR method, while the needle is inserted at a 90-degree angle, deep pressure will be applied to the muscle, then rapidly released to create a snapping motion that facilitates the injection. This technique relies on rapid muscle relaxation rather than needle movement by the dominant hand.
  Interventions: Other: TPR method
- Z-track method (Experimental): Intervention Type: Intramuscular drug administration with Z-track method Intervention Name: Diclofenac Sodium Z-track method, the skin will be pulled laterally by 2.5-3.5 cm before needle insertion at a 90-degree angle. After aspiration and injection, the needle will be withdrawn and the skin released immediately.
  Interventions: Other: Z-track method

INTERVENTIONS:
Other: Z-track method — Z-track method, the skin will be pulled laterally by 2.5-3.5 cm before needle insertion at a 90-degree angle. After aspiration and injection, the needle will be withdrawn and the skin released immediately.
  Arms: Z-track method
Other: TPR method — TPR method, while the needle is inserted at a 90-degree angle, deep pressure will be applied to the muscle, then rapidly released to create a snapping motion that facilitates the injection. This technique relies on rapid muscle relaxation rather than needle movement by the dominant hand.
  Arms: TPR (traction-pressure-release) technique

SUMMARY:
This randomized, triple-blind clinical trial compares the effectiveness of Z-track and TPR (traction-pressure-release) techniques in reducing pain and medication leakage during ventrogluteal intramuscular injections. Pain is measured using VAS, and leakage is assessed with a millimeter scale. The study aims to identify a more efficient, less painful injection method.

DETAILED DESCRIPTION:
Introduction: Intramuscular (IM) injections are widely used for delivering medications due to their high bioavailability and quick absorption. However, they can cause significant local complications, especially pain, which may affect patient compliance. Various non-pharmacological techniques have been developed to reduce injection pain, including the Z-track method and the more recent TPR (traction-pressure-release) technique, based on the gate control theory of pain. While both aim to minimize pain, TPR has shown promise but lacks research regarding its effect on drug leakage.

Objective: The study aims to compare the effectiveness of TPR and Z-track techniques in reducing pain and drug leakage during IM injections in the ventrogluteal site.

Method: This study is a triple-blind, randomized, two-group clinical trial with a parallel design. A total of 76 patients aged 16-40, prescribed with intramuscular diclofenac sodium, will be recruited. Each participant will receive both techniques-TPR and Z-track-in randomly assigned ventrogluteal muscles. Pain intensity will be measured using a Visual Analog Scale (VAS), and drug leakage will be assessed using millimetric paper and a ruler. All injections will be administered by the same nurse, and evaluation will be performed by blinded assessors.

Conclusion: This research seeks to provide evidence on the efficacy of the TPR technique as a potentially time- and cost-effective alternative to Z-track, particularly in minimizing injection-related pain and leakage, thereby improving patient comfort and treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-40
* Prescribed diclofenac sodium
* No communication impairments
* Healthy ventrogluteal muscles without sensory issues

Exclusion Criteria:

* Wounds, redness, bruising, tenderness, or stiffness at the injection site
* Injection in the past 2 weeks
* Neuropathy or other medical conditions
* BMI below 15 or above 35

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
Pain with visual analog scale | Within 5 minutes after intramuscular injection
  Pain intensity measured with the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicate greater pain.

SECONDARY OUTCOMES:
Drug leakage | Time Frame: Immediately after injection (within 1 minute)Description: Drug leakage will be observed immediately after intramuscular injection by checking the injection site for any visible medication leakage.
  millimeter ruler to assess medication leakage

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda Kazanç, Phd, Study Director — but no location
Locations (2):
- Turkey (Türkiye) (2):
  - Sivas Numune Hospital, Sivas
  - Sivas State Hospital, Sivas

IPD SHARING:
Plan to Share IPD: No
I would like to share the research after it is completed.